CLINICAL TRIAL: NCT03780699
Title: Hysteroscopic Evaluation of Cesarean Scar Defect Features & Its Correlation With Women Complaints
Brief Title: Hysteroscopic Evaluation of Cesarean Scar Defect
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, Principal Investigator, Ain Shams University
Other Study IDs: Ain Shams University H
Record Dates: First submitted 2018-12-16; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cesarean Scar Defect

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Diagnostic hysteroscopic examination — The hysteroscopic criteria of the cesarean scar defect will be observed with comment on different niche features

SUMMARY:
The aim of this study is to identify hysteroscopic findings of cesarean scar defect in women underwent at least one prior cesarean section and its relation to any of the different un explained gynecological presentations.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 35 years.
2. Had at least one prior cesarean section

Exclusion Criteria:

1. History of uterine surgery that could change the cavity anatomy.
2. Uterine Abnormalities as submucous fibroid, endometrial or endocervical Polyps.
3. Recent intra-uterine contraceptive device (IUCD) in place.
4. Known history of endometriosis

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be carried on 200 patients with cesarean scar defect recruited from Early Cancer Detection Unit.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
cesarean section scar defect shapes | at least six months after CS
  different shapes of CS defect and its relation to post menstrual spotting

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Abbassya, Egypt

IPD SHARING:
Plan to Share IPD: No